CLINICAL TRIAL: NCT06950905
Title: Effectiveness of a Contemplative Practice on Psychological Well-Being, Self-Deconstruction, Body Image, Body Acceptance, and Compassion in Women
Brief Title: Contemplative Practice for Well-being and Self-Deconstruction in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI25/008
Record Dates: First submitted 2025-04-02; First posted 2025-04-30 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Mental Health; Self Concept; Body Dissatisfaction; Compassion; Self-Perception; Mindfulness Meditation; Meditation; Psychological Well-being
Keywords: Feeding Your Demons; Self-Deconstruction; Selflessness; Contemplative Practices; Meditation; Compassion; Body Image; Women's Mental Health; Randomized Controlled Trial (RCT); mindfulness; psychological well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Feeding Your Demons practice (Experimental): The experimental group will engage in a "Feeding Your Demons" contemplative practice involving repeated sessions (30-60 minutes each).
  The practice follows this structured protocol across sessions:
  Preparation: Preparation: Comfortable sitting posture in a chair, with an empty chair in front.
  Theme/Visualization: Identify a challenge (e.g., self-criticism, body dissatisfaction), observe bodily sensations, personify as a "demon" (note traits).
  Dialogue: Shift chairs, embody the demon, answer: What do you want? Need? How will you feel when fulfilled?
  Transformation: Return, dissolve demon into "nectar" (embodying its need), feed until it becomes an ally.
  Ally Engagement: Note ally's traits, ask: How will you help/protect? What promise? How to access you? Briefly embody ally.
  Closure: Ally dissolves into participant; and both dissolves and rest in present-moment awareness.
  Interventions: Behavioral: Feeding your demons practice
- Mindfulness Meditation condition (Active Comparator): The control group will engage in a mindfulness meditation intervention involving repeated sessions (30-60 minutes each). The practice follows this structured protocol across sessions:
  Preparation and Posture: Participants adopt a comfortable seated position with an upright spinal alignment.
  Breath Awareness: Sustained attention is directed toward natural respiratory rhythms without deliberate modulation.
  Body Scan: Systematic observation of somatic states (e.g., tension or relaxation) across distinct anatomical regions.
  Observation of Thoughts and Emotions: Transient cognitive and affective phenomena are acknowledged with non-judgmental detachment, avoiding engagement.
  Closure: Each session concludes with a return to breath-centered focus and gradual reorientation to the external environment.
  Interventions: Behavioral: Mindfulness practice

INTERVENTIONS:
Behavioral: Feeding your demons practice — The Feeding Your Demons (FYD) is a contemplative practice based on the Tibetan Buddhist tradition, adapted in a secular form. The intervention is online and lasts a total of 8 weeks. During this period, participants will engage in weekly home practice of the FYD method using guided audio. The intervention includes 3 expert-facilitated sessions: an initial individual session, a group session at week 4, and a final group session at week 8.
  Other Names: Feeding your demons; FYD
  Arms: Feeding Your Demons practice
Behavioral: Mindfulness practice — The control group will undergo an online mindfulness meditation intervention, lasting a total of 8 weeks. It includes 3 expert-facilitated sessions: an initial individual session, a group session at week 4, and a final group session at week 8. Participants will engage in weekly home practice of mindfulness meditation using guided audio.
  Other Names: Mindfulness; Mindfulness meditation; Attentional meditation
  Arms: Mindfulness Meditation condition

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of a contemplative practice called Feeding Your Demons (FYD), based on a secular adaptation of Tibetan Buddhism, in improving psychological well-being, body image, body acceptance, compassion, and self-deconstruction in adult women. Participants will be randomly assigned to either FYD or an active control group practicing mindfulness meditation. Psychological variables will be assessed before and after the intervention, and at a six-month follow-up. Additionally, a qualitative exploration will be conducted through interviews with a subgroup of participants.

DETAILED DESCRIPTION:
Feeding Your Demons (FYD) is a secular contemplative practice inspired by the Tibetan Buddhist tradition, integrating elements of mindfulness, compassion, and symbolic visualization. The practice offers a guided process through which individuals face internal difficulties-referred to as "demons"-and transform them through acceptance and self-compassion.

This study aims to evaluate the effectiveness of FYD compared to a mindfulness meditation intervention. It is a randomized controlled trial (RCT) with two parallel groups. A total of 122 adult women will participate. Participants will be randomly assigned to either the FYD group or the control group. Both interventions will be delivered online over eight weeks.

Variables assessed include psychological well-being, body image, body acceptance, mindfulness, compassion, and self-deconstruction. Assessments will be conducted before and after the intervention, and at a six-month follow-up.

Statistical analyses will include intra- and intergroup comparisons using repeated measures analysis of variance. Parametric or non-parametric tests will be applied depending on the assumptions met. Relationships between variables will also be analyzed through correlations. Effect sizes will be calculated to estimate the magnitude of observed changes. The significance level will be set at p < .05, with a 95% confidence interval.

This study adopts a mixed-methods approach, combining quantitative assessments with qualitative interviews conducted with a subgroup of participants. Although the data are collected complementarily, their analysis and dissemination may be conducted separately or integratively, depending on the specific goals of each research phase.

ELIGIBILITY:
Inclusion Criteria:

* Sex assigned female at birth and self-identifies as a woman
* Aged between 30 and 60 years
* Spanish nationality, or residency in Spain for more than 5 years
* Fluent in Spanish
* At least one month of experience with meditation or mindfulness practices, with a regular practice of more than 15 minutes per session
* Provides informed consent

Exclusion Criteria:

* Indicators of eating disorders (ED) or mental health deterioration, determined by the following cut-off points: SCOFF ≥ 2 and PHQ-9 ≥ 10
* Formal diagnosis of an eating disorder or any psychiatric condition
* Substance use disorder
* History of neurological disease diagnosis
* Participant's decision to withdraw from the study at any point

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only individuals who were assigned female at birth and who currently self-identify as women are eligible to participate in the study. This criterion ensures alignment with the study's focus on female embodiment, body image, and self-related perception in adult women.
Enrollment: 122 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Delusion of Me Index (DoM) | From baseline to 6-month follow-up
  The primary outcome will be the change in self-related perception from baseline to 6-month follow-up after randomisation. This includes changes in acceptance, decentering, and non-attachment. Participants will complete this measure at three time points: baseline (week 0), post-intervention (week 8), and 6-month follow-up.
Nondual Awareness Dimensional Assessment (NADA) | From baseline to 6-month follow-up
  The primary outcome will be the change in self-related perception from baseline to 6-month follow-up after randomisation. This outcome includes changes in nondual awareness. Participants will complete this measure at three time points: baseline (week 0), post-intervention (week 8), and 6-month follow-up.
Body Appreciation Scale-2 (BAS-2) | From baseline to 6-month follow-up
  The second primary outcome will be the change in body image from baseline to 6-month follow-up after randomisation. This includes improvements in positive body image, specifically body appreciation. Participants will complete this measure at three time points: baseline (week 0), post-intervention (week 8), and 6-month follow-up.
Body Shape Questionnaire-10 (BSQ-10) | From baseline to 6-month follow-up
  The second primary outcome will be the change in body image from baseline to 6-month follow-up after randomisation. This includes reductions in negative body image, specifically body dissatisfaction. Participants will complete this measure at three time points: baseline (week 0), post-intervention (week 8), and 6-month follow-up.

SECONDARY OUTCOMES:
Pemberton Happiness Index (PHI) | From baseline to 6-month follow-up
  Change in Psychological Well- Being
SOCS-S Sussex-Oxford Self- Compassion Scale | From baseline to 6-month follow-up
  Change in Self - Compassion
Five Facet Mindfulness Questionnaire (FFMQ). | From baseline to 6-month follow-up
  Change in Mindfulness
Body Image Acceptance and Action Questionnaire (BI-AAQ-5). | From baseline to 6-month follow-up
  Change in Body Acceptance
Sussex- Oxford Compassion Scale (SOCS - O) | From baseline to 6-month follow-up
  Change in Compassion (for others)
Multidimensional Assessment of Interoceptive Awareness (MAIA) | From baseline to 6-month follow-up
  Change in Interoceptive Awareness

OTHER OUTCOMES:
Participant Age | At baseline
  Age of participants, measured in years.
Place of Residence | At baseline
  The place of residence (e.g., community or city) of participants will be recorded at baseline.
Education Level | At baseline
  Participants will report their highest completed education level at baseline.
Employment Status | At baseline
  Employment status (e.g., employed, unemployed, student) will be collected at baseline.
Prior Meditation Experience | At baseline
  Participants will report whether they have prior meditation experience (yes/no) and, if applicable, the number of months or years of practice.Additionally, they will indicate the type of meditation practice previously performed (e.g., mindfulness, compassion, other).
Number of Meditation Session | During the 8-week intervention
  Participants will indicate the sequential number of each formal meditation session completed during the 8-week intervention (e.g., Session 1, Session 2, Session 3).
Perceived Quality of Meditation Practice | During the 8-week intervention
  After each formal meditation session, participants will rate the perceived quality of their practice on a scale from 0 (very poor) to 10 (excellent).
Self-reported Affective State after Practice | During the 8-week intervention
  Participants will rate their affective state immediately after each formal meditation session on a scale from 0 (very negative) to 10 (very positive).
Qualitative phenomenological exploration | From baseline to post-intervention (8 weeks after baseline)
  Semi-structured micro-phenomenological interviews will be conducted at baseline and immediately after the 8-week intervention to explore participants' lived experience related to self-perception, embodiment, and contemplative transformation. These data are exploratory and will not be included in inferential statistical analyses.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Department of Psychiatry. Miguel Servet University Hospital, Zaragoza, Zaragoza
  - University of Zaragoza, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No